CLINICAL TRIAL: NCT01690221
Title: A Phase 3B, Randomized, Double-Blind, Placebo-Controlled, Parallel-Treatment Group, Multicenter Efficacy and Safety Study of Topical Diltiazem Hydrochloride 2% Cream in Subjects With Anal Fissure
Brief Title: Efficacy and Safety Study With Diltiazem Hydrochloride Cream to Treat Anal Fissures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEN307-AF-001
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Anal Fissures
Keywords: Anal; Fissure; Pain
MeSH Terms: conditions — Pain | interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VEN 307 (Experimental): diltiazem hydrochloride 2% cream
  Interventions: Drug: VEN 307
- Placebo (Placebo Comparator): Placebo Cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VEN 307 — VEN307 applied three times a day, in and around the anus, for 28 days.
  Other Names: diltiazem hydrochloride 2% cream
  Arms: VEN 307
Drug: Placebo — Placebo cream applied three times a day, in and around the anus, for 28 days.
  Other Names: Placebo cream
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the study drug, VEN307 (diltiazem hydrochloride cream) is safe and to see if it will help with treatment of pain associated with anal fissures.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of diltiazem hydrochloride cream on reduction of worst anal fissure (AF)-related pain associated with or following defecation when administered three times a day (TID) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 18 to ≤ 75 years.
2. Subjects with evidence of a circumscribed fissure, with induration at the edges.
3. Subjects with AF-related pain associated with or following defecation occurring at least 2 times a week for at least 28 days prior to signing the informed consent form (ICF).
4. AF-related pain associated with or following defecation of at least 5 on an 11-point numerical rating score scale (NRS) at the last defecation prior to signing the ICF (0 being no pain; 10 being the worst possible pain).
5. Average AF-related pain associated with or following defecation of at least 5 on an 11-point NRS during the last 3 days in which subject had a defecation during the 7 days prior to randomization.
6. Any female of non-childbearing potential, including any female who: a) has had a hysterectomy, b) has had a bilateral oophorectomy, c) has had a bilateral tubal ligation or d) is post menopausal (demonstration of total cessation of menses for ≥ 1 year from the date of screening visit).
7. Females of child bearing potential who agree to use at least one form of contraception (may be a barrier method), during the full duration of the study.
8. Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
9. Capable of using the IVRS and able to adequately communicate comprehension of the IVRS questions to the investigator.
10. Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

1. Unwilling to have visual or medical examination of the AF.
2. More than 1 AF.
3. Subjects with AF associated with or caused by other conditions, including but not limited to: drug-induced, trauma, HIV infection, fistula-in-ano, inflammatory bowel disease, perianal sepsis or malignancy.
4. Unwilling to stop all other concomitant topical preparations applied in and around the anus from signing of ICF through Day 29 of the study.
5. Use of glyceryl trinitrate (GTN) ointment for 7 days (continuous or not) in the 28 days prior to signing the ICF.
6. Unwilling to discontinue use of sitz baths for up to 4 hours after each application of investigational product from signing of ICF to end of study.
7. Unwilling to discontinue use of anesthetics from signing the ICF to end of study.
8. Subfissure injection of botulinum toxin in the 3 months prior to signing the ICF.
9. Known sensitivity to investigational product(s) or calcium channel blockers.
10. Previous treatment with diltiazem hydrochloride cream or any other topical calcium channel blockers.
11. Active treatment with anti-viral therapies for HIV (e.g. indinavir, nelfinivir, ritonavir).
12. Treatment with any of the following medications within 14 days prior to signing the ICF:

    * Amitriptyline
    * Benzodiazepines
    * β-adrenoceptor antagonists (Beta-Blockers)
    * Buspirone
    * Calcium channel blockers
    * Carbamazepine
    * Cimetidine
    * Cyclosporin
    * Digoxin
    * Investigational agents
    * Lovastatin
    * Opioids
    * Pregabalin
    * Quinidine
    * Rifampin
13. Following concomitant disease state:

    * Sick sinus syndrome except in the presence of a functioning ventricular pacemaker.
    * Second-or third-degree AV block except in the presence of a functioning ventricular pacemaker.
    * Hypotension (less than 90 mm Hg systolic).
    * Acute myocardial infarction and pulmonary congestion documented by x-ray.
    * History of bipolar disorder, psychosis, schizophrenia, mania, suicide attempt or suicidal ideation, or any other significant psychiatric illness (with the exception of intermittent anxiety) per investigator judgment.
    * History of clinically significant renal disease per investigator judgment.
    * History of clinically significant Alzheimer's or Parkinson's disease per investigator judgment.
    * History of clinically significant hepatic disease per investigator judgment.
    * Current infection treated with a macrolide antibiotic.
    * Clinical evidence or history of fecal incontinence.
    * Clinical evidence or history of anal fistula.
    * Clinical evidence or history of anal abscess.
    * History of inflammatory bowel disease (e.g. Crohn's disease, Ulcerative Colitis).
    * History of any prior anal or rectal surgery including but not limited to: lateral sphincterotomy and anal stretch (with the exception of hemorrhoidal banding and laser surgery).
    * Grade 4 hemorrhoids.
    * Chronic constipation.
14. History of radiation therapy to the pelvis.
15. Fixed anal stenosis/fibrosis.
16. Major organ transplant.
17. Any clinically significant laboratory abnormalities during screening per investigator judgment.
18. Body Mass Index (BMI) > 40 kg/m2
19. Malignancy within 5 years prior to randomization (with the exception of treated basal cell/squamous cell carcinoma of the skin).
20. Any disease or prior/planned surgery that may interfere with the subject successfully completing the study.
21. Currently using narcotic(s).
22. Breast-feeding females.
23. Employees, family members, or students of the investigator or clinical site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline (average NRS during the last 3 days in which subject had a defecation during the 7 day screening period) in average of worst AF-related pain associated with or following defecation for Days 22-28 (Week 4). | 28 days

CONTACTS AND LOCATIONS:
Locations (103):
- United States (103):
  - The Crawford Clinic, Anniston, Alabama
  - Surgical Association of Mobile, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama
  - Montgomery Women's Health Association, PC, Montgomery, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - UC San Diego, La Jolla, California
  - Alliance Research Centers, Laguna Hills, California
  - Axis Clinical Trials, Los Angeles, California
  - Cedars Sinai, Los Angeles, California
  - Gastrointestinal Biosciences, Los Angeles, California
  - University of California - Irvine Medical Center, Orange, California
  - Digestive Care Associated, A Medical Corporation, San Carlos, California
  - West Coast Clinical Research, Tarzana, California
  - Rocky Mountain Clinical Research, LLC, Denver, Colorado
  - Colorado Research Works, Pueblo, Colorado
  - Rocky Mountain Clinical Research, LLC, Thornton, Colorado
  - Connecticut Clinical Research Foundation CT Gastroenterology Institute At Bristol Hospital, Bristol, Connecticut
  - Washington Hospital Center - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Innovative Medical Research of South Florida, Aventura, Florida
  - South Lake Pain Institute, Clermont, Florida
  - Private Practice, Hollywood, Florida
  - Advance Medical Research Center, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Akta Medika, Miami Beach, Florida
  - Gastroenterology Group of Naples, PA, Naples, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Private Practice, Pembroke Pines, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - University of South Florida, South Campus, Tampa, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Atlanta Center for Gastroenterology, Decatur, Georgia
  - Gastrointestinal Specialist of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Consultants, Suwanee, Georgia
  - NCH Medical Group, Arlington Heights, Illinois
  - North Shore University Health System, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Kendrick Regional Medical Center, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Monroe, Louisiana
  - Ochsner, New Orleans, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center Department of Surgery, Springfield, Massachusetts
  - Center for Digestive Health, Troy, Michigan
  - CRC of Jackson, Jackson, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Midwest Center for Clinical Research, Lee's Summit, Missouri
  - Colon and Rectal Surgery, Inc, Omaha, Nebraska
  - Impact Clinical Trials, Las Vegas, Nevada
  - Gastroenterology Group & Endoscopy Center of South NJ (GGSJ), Vineland, New Jersey
  - C&R Surgical Assoc of South Jersey, Voorhees Township, New Jersey
  - Life Medi-Research and Management, Brooklyn, New York
  - HCCA Clinical Research Solutions, New York, New York
  - Manhattan Surgical Associates, LLP, New York, New York
  - Colorectal Associates of NY, New York, New York
  - Medical Research Associates of New York (New York Gastroenterology Associates, LLP), New York, New York
  - Premier Medical Group, Poughkeepsie, New York
  - Medispect, Boone, North Carolina
  - Duke University, Durham, North Carolina
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - University of North Carolina, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Gastroenterology, Inc., Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Institute of Pain Research, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - The Corvallis Clinic, Clinical Research Center, Corvallis, Oregon
  - Westover Heights Clinic, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - West Penn Allegheny Health System, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Drexel Univ College of Medicine, Philadelphia, Pennsylvania
  - Temple University Physicians, Jeanes Hospital, Philadelphia, Pennsylvania
  - Pain Specialists of Charleston, North Charleston, South Carolina
  - Gastroenterology Associates of Orangeburg, PA, Orangeburg, South Carolina
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - Vanderbilt Univ Dept of Colon and Rectal Surgery, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Research Concepts, GP LLC, Houston, Texas
  - University of TX Affiliated Hospitals, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Houston Digestive Disease Clinic, Houston, Texas
  - ColoProctology Associates, Seabrook, Texas
  - University of Utah HSC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Jefferson Surgical Clinic, Roanoke, Virginia
  - NW Gastroenterology, Bellevue, Washington
  - Digestive Disease Institute, Virginia Mason Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Medical College of Wisconsin Department of Surgery, Milwaukee, Wisconsin